CLINICAL TRIAL: NCT03230253
Title: Effects and Mechanism of Two Hybrid Exercise-cognitive Trainings in Mild Ischemic Stroke With Cognitive Decline: fMRI for Brain Plasticity, and Biomarker and Behavioral Analysis
Brief Title: Effects and Mechanism of Two Hybrid Exercise-cognitive Trainings in Mild Ischemic Stroke With Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20170040
Record Dates: First submitted 2017-07-18; First posted 2017-07-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Stroke Patients With Cognitive Decline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequential training group (Experimental): Exercise training for 30 minutes followed by 30 minutes of cognitive-based intervention
  Interventions: Behavioral: Sequential training
- Dual training group (Experimental): Exercise training simultaneously combined cognitive-based intervention for 60 minutes
  Interventions: Behavioral: Dual training
- Control training group (Active Comparator): non-aerobic exercise (e.g., stretch, range of motion exercise...) and unstructured cognitive rehabilitation programs (e.g., reading newspapers, playing board games...) for 60 minutes
  Interventions: Behavioral: Control training

INTERVENTIONS:
Behavioral: Sequential training — The participant will cycle on a stationary bike for 30 minutes, which includes a 3-min warm-up phase followed by the aerobic training components (25 minutes), then a 2-min cool-down phase. The target heart rate during the aerobic training phase will be 40 to 70% of maximal heart rate (HRmax). After cycling, the participant will engage in a 30-minute of computer-based cognitive training program using BrainHQ (Posit Science Inc., San Francisco, CA, USA). The following are the areas of training: visuospatial processing, attention, memory, language, and logical thinking.
  Arms: Sequential training group
Behavioral: Dual training — The dual-task training group will cycling concurrently with the computer-based cognitive training. The training principle of cycling and cognitive training is similar to the SEQ group; however, the training intensity will be adjusted according to each participant's ability.
  Arms: Dual training group
Behavioral: Control training — The control participants will receive 60 minutes of health-related rehabilitation programs which involves non-aerobic physical exercise (e.g., muscle stretching, range of motion exercises, relaxation techniques) and unstructured cognitive related rehabilitation programs (e.g., watch health-related videos or read newspapers or magazines and then answer the content-related questions raised by the therapist).
  Arms: Control training group

SUMMARY:
The purposes are to: (1) examine and compare the effects of two hybrid interventions on brain plasticity, physiological biomarkers and behavioral outcomes, including cognitive and physical functions, from pre- to post-training; (2) understand the neural mechanisms of cognitive recovery following two hybrid interventions using the functional magnetic resonance imaging (fMRI); (3) examine the long-term benefits of the two hybrid therapies; (4) to identify the correlations between brain activity, biomarkers and behavioral measures.

DETAILED DESCRIPTION:
Cognitive decline after stroke is highly associated with functional disability. Empirical evidence shows that exercise combined cognitive training may induce neuroplastic changes that modulate cognitive function. However, it is unclear whether hybridized exercise-cognitive trainings can facilitate cortical activity and physiological outcome measures and further influence on the cognitive function after stroke. We aim to investigate the effects of two hybridized exercise-cognitive trainings on brain plasticity, physiological biomarkers and behavioral outcomes in stroke survivors with cognitive decline. This study is a single-blind randomized controlled trial. A target sample size of 75 participants will be recruited. Stroke survivors with mild cognitive decline will be stratified by Mini-Mental State Examination scores and then randomized 1:1:1 to sequential exercise-cognitive training, dual-task exercise-cognitive training or control groups. All groups will undergo trainings 60 min/day, 3 days/week, for a total of 12 weeks. The primary outcome is the resting-state functional connectivity and neural activation in the frontal, parietal and occipital lobes in functional magnetic resonance imaging. Secondary outcomes include physiological biomarkers, cognitive functions, physical function, daily functions and quality of life.

This study may differentiate the effects of two hybridized trainings on cognitive function and health-related conditions and detect appropriate neurological and physiological indices to predict training effects. This study capitalizes on the groundwork for non-pharmacological intervention of cognitive decline after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke occurring at least 6 months prior to enrollment
2. Age range from 20 to 80 years
3. MMSE score < 28 or MoCA<25
4. Able to follow the study instruction
5. Adequate cardiopulmonary function to perform aerobic exercise
6. Able to walk with or without assistive devices

Exclusion Criteria:

1. Unstable medical history (e.g., recent myocardial infarction) that might limit participation
2. Concomitant with other neurological disorders (e.g., Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis)
3. Current participation in another interventional trial
4. Any contraindication to MRI (metallic implants, claustrophobia, seizure, pacemakers, et al)
5. Pregnant woman

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
fMRI (change is being assessed) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months).
  Resting-state functional connectivity and neural activation in the frontal, parietal and occipital lobes

SECONDARY OUTCOMES:
Serum BDNF level | Baseline, posttest (an expected average of 3 months)
  Up-regulation of neurotrophic and vascular growth factors
Antioxidative marker | Baseline, posttest (an expected average of 3 months)]
  Antioxidative markers will be used to reflect the changes on oxidative stress. In particular, we will be analyzing the total antioxidant capacity (TAC).
Glucose indicator | Baseline, posttest (an expected average of 3 months)
  HbA1C level will be tested to investigate the relationships between blood glucose level and aerobic exercise
Plasma lipid level | Baseline, posttest (an expected average of 3 months)
  The cholesterol ratio (total cholesterol divided by high-density lipid) will be evaluated to reflect the lipid level in the blood
Montreal Cognitive Assessment (MoCA) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The MoCA will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30
Wechsler Memory Scale - Third Edition (WMS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The WMS-III is a standardized and reliable neuropsychological examination tool designed to evaluate visuospatial and memory functions
Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The WAIS-III is developed to measure an individual's intelligence level. It includes tests that evaluate cognitive functions in verbal comprehension, working memory, perceptual organization, and processing speed
Useful Field of View (UFOV) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The UFOV assessment is a computer-based visual test containing three subtests: visuomotor processing speed, divided attention, and selective attention.
Stroop Color-Word test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Stroop Color-Word assesses the abilities of selective attention, inhibition and executive function. The participants will be tested under congruent and incongruent conditions.
Dual-task test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The dual-task test evaluates the ability to shift attention between one task and another. Participants will perform the box and block test (BBT) while doing secondary cognitive tasks while sitting. Participants will perform BBT by affected and less affected hand.
Time up and go test (TUG) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The TUG assesses the dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down.
Six-minute walk test (6MWT) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The 6MWT measures the maximum distance walked over 6 minutes, which assess the endurance and mobility level of the participants. The participants could rest as needed during the course of the test.
International Physical Activity Questionnaires (IPAQ) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The IPAQ is an international measure of health-related physical activity.
Fugl-Meyer Assessment (FMA) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The 33-item upper limb subscale of the FMA will be used to assess motor impairments.
Rivermead Mobility Index (RMI) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The RMI evaluates the participant's bed mobility, postural transfers and walking ability. It contains a 15-item scale which includes 14 questions and one direct observation, with a total of score of 15.
Muscle strength | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Accelerometers will be used to provide an objective measure of the amount of arm movements in real-life situations. The participants will be asked to wear an Actigraphy activity monitor.
Mobility level | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Accelerometers will be used to provide an objective measure of the amount of arm movements in real-life situations. The participants will be asked to wear an Actigraphy activity monitor.
Functional Independence Measure (FIM) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The FIM assesses the dependence level of individuals with stroke to perform 18 activities (13 motor and five cognitive tasks) in daily living. The score ranges from 18 to 126 and higher scores demonstrate greater independent participation in daily activities.
Lawton Instrumental Activities of Daily Living Scale (Lawton LADL) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Lawton IADL scale assesses independent living skills, such as shopping or managing finances.
Stroke Impact Scale (SIS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The SIS 3.0 will be used to evaluate health-related quality of life for patients with stroke. The SIS assesses eight domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, and participation/role function) with 59 test items.
Caregiver Burden Scale (CB scale) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  B scale evaluates the burden of the primary caregiver of the participants. Lessening the burden of caregivers after the intervention may significantly improve the quality of life for patients with stroke and their family.
EuroQol-5D questionnaire (EQ-5D) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The quality of life will be assessed by the EQ-5D questionnaire which comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Kaohsiung Municipal Siaogang Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Yeh TT, Chang KC, Wang JJ, Lin WC, Wu CY. Neuroplastic Changes Associated With Hybrid Exercise-Cognitive Training in Stroke Survivors With Mild Cognitive Decline: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2023 Sep;37(9):662-673. doi: 10.1177/15459683231200220. PMID 37750660
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186